CLINICAL TRIAL: NCT00714701
Title: Screening for Early Pancreatic Neoplasia (Cancer of the Pancreas Screening or CAPS4 Study)
Acronym: CAPS4
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The V Foundation for Cancer Research (Other); ChiRhoClin, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: J0139 00-04-14-10; J0139; NCT00084357 (obsolete NCT alias)
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Early Pancreatic Neoplasia; Familial Pancreatic Neoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, pancreatic juices
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- High Risk Group 1: familial Peutz-Jeghers syndrome
- High Risk Group 2: familial pancreatic cancer relatives
- High Risk Group 3: germline mutation carriers BRCA1, BRCA2, PRSS, PALB2, p16
- High Risk Group 4: young-onset pancreatic cancer relative
- High Risk Group 5: both parents affected
- Control 1: negative controls
- Control 2: chronic pancreatitis
- Control 3: pancreatic cancer
- Control 4: intraductal papillary mucinous neoplasm (IPMN)

SUMMARY:
CAPS4 is a study at Johns Hopkins Hospital to study the diagnosis and long-term outcomes of screening patients with an increased inherited risk for pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is a deadly disease and the only hope for improvement of survival is early detection. Certain genetic syndromes are associated with a high risk of pancreatic cancer and screening for pancreatic cancer has become a relatively new strategy for familial pancreatic cancer. . Our pancreatic cancer research group at Johns Hopkins and others have shown that screening with EUS and/or abdominal imaging tests such as CT/MRI can detect a relatively high number of significant pancreatic neoplasms (7-18%) in asymptomatic high risk individuals with an inherited predisposition for pancreatic ductal adenocarcinoma This is a clinical, early detection translational study that will directly influence patient care. This long term study follows the successful completion of single center Cancer of the Pancreas (CAPS) 1 and CAPS 2 studies at Johns Hopkins, and the ongoing CAPS 3 multicenter study. GENERAL AIM: This is a study that aims to evaluate the diagnostic yield, quality of life, and clinical outcomes of a clinical screening and surveillance program for individuals at-risk for pancreatic cancer and to validate a candidate panel of biomarkers for early detection of pancreatic neoplasia. The 3 specific groups to be screened and followed are individuals from familial pancreatic cancer kindreds (who have 2 or more affected relatives and have an estimated risk 16-57 times that of controls), patients with familial Peutz-Jeghers syndrome, patients with a known BRCA-2, BRCA-1, PALB2, PRSS or p16 germline mutation.

ELIGIBILITY:
Inclusion Criteria:

1. High Risk Group 1 (familial Peutz-Jeghers syndrome):

   1. At least 30 years old and <100 years old, and
   2. at least 2 of 3 criteria diagnostic of Peutz-Jeghers syndrome (characteristic intestinal hamartomatous polyps, mucocutaneous melanin deposition, or family history of Peutz-Jeghers syndrome)
   3. known STK-11 gene mutation carrier
2. High Risk Group 2 (familial pancreatic cancer relatives):

   1. > 50 years old or 10 years younger than the age of youngest relative with pancreatic cancer, and < 80 years old
   2. come from a family with 2 or more members with a history of pancreatic cancer (2 of which have a first-degree relationship consistent with familial pancreatic cancer), and
   3. have a first-degree relationship with at least one of the relatives with pancreatic cancer.

   If there are 2 or more affected blood relatives, at least 1 must be a first-degree relative of the individual being screened
3. High Risk Group 3 (germline mutation carriers):

   1. > 40 years old or 10 years younger than the age of the youngest relative with pancreatic cancer, and< 80 years old
   2. patient is carrier of a known BRCA1, BRCA2, PALB2, or FAMMM (p16/CDKN2A) mutation, and there is > 1 pancreatic cancer in the family, one of whom is a first- or second-degree relative of the subject to be screened.
   3. Hereditary pancreatitis syndrome
4. High Risk Group 4 (young-onset pancreatic cancer relative):

   1. > 50 years old or 10 years younger than the age of youngest relative with pancreatic cancer, and < 80 years old
   2. have a first-degree relationship with at least one relative with young-onset pancreatic cancer ( age of onset < 50 years)
5. High risk group 5 (both parents affected)

   1. > 50 years old or 10 years younger than the age of the youngest relative with pancreatic cancer, and< 80 years old
   2. two parents affected by pancreatic cancer
6. Control 1 (Negative Controls):

   1. are undergoing EUS and/or ERCP for non-pancreatic indications as part of their standard medical care, and
   2. have no clinical or radiologic suspicion of pancreatic disease (chronic pancreatitis or pancreatic cancer)
7. Control 2 (Chronic Pancreatitis)

   1. are undergoing EUS and/or ERCP for evaluation and/or treatment of suspected or proven chronic pancreatitis as part of their standard medical care, and,
   2. have no clinical or radiologic suspicion of pancreatic cancer
8. Control 3 (Pancreatic Cancer)

   a. are undergoing EUS and/or ERCP for evaluation and/or treatment of suspected or proven pancreatic ductal adenocarcinoma (based on clinical and radiologic evidence)
9. Control 4 (Intraductal Papillary Mucinous Neoplasm or IPMN) a. are undergoing EUS and/or ERCP for evaluation and/or treatment of suspected or proven pancreatic cancer precursor, intraductal papillary mucinous neoplasm (based on clinical presentation and radiologic or prior EUS or radiologic evidence of a dilated main pancreatic duct and/or pancreatic cystic lesion communicating with the pancreatic ductal system)

Additional requirements for eligible high risk patients: i) All persons with known genetic mutation must have proof of mutation status. Those who had research-related genetic testing must have confirmation by a clinical CLIA-certified laboratory. ii) A good faith attempt should be made to confirm pancreatic cancers in the family members via registration in a pancreatic cancer registry iii) The affected first degree relative of the person being screened must be confirmed by medical record or death certificate.

All control patients must be > 18 and < 80 years old and no personal or family history of pancreatic cancer or a germline mutation linked to pancreatic cancer.

Exclusion Criteria:

Patients will be excluded if they have any of the following:

1. medical comorbidities or coagulopathy that contraindicate endoscopy,
2. Karnosfky performance status of < 60,
3. had partial or complete resection of their pancreas
4. had a partial or complete gastrectomy with Billroth or Roux-en-Y anastomosis
5. a stricture or obstruction in the upper GI tract that does not allow passage of the echoendoscope
6. life expectancy less than 5 years due to coexisting advanced cancer or AIDS.
7. inability to provide informed consent
8. pregnant patient
9. history of pancreatic cancer,
10. suspicion of pancreatic neoplasia based on clinical history (weight loss, unexplained abdominal pain), physical examination (obstructive jaundice, cachexia), laboratory tests (cholestastic liver function tests, markedly elevated CA19-9), and/or imaging studies (pancreatic mass or cyst, dilated pancreatic and/or bile duct);
11. there is no interest in undergoing treatment of pancreatic neoplasm(s) detected by screening.
12. history of chronic kidney disease, serum creatinine > 2.0 mg/dl or estimated glomerulofiltration rate (eGFR) < 30 ml/min, ongoing acute renal failure, cirrhosis of the liver, chronic hepatitis (The estimated glomerulfiltration rate (eGFR) will be calculated based on age, race, and serum creatinine, using the on-line calculator at nephron.com).
13. history of dementia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: asymptomatic high risk patients
Sampling Method: Probability Sample
Enrollment: 631 (Actual)
Dates: Start 2008-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
This clinical study will assess the diagnostic yield of a clinical screening program for early pancreatic neoplasia in high risk individuals. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Irene F. Canto, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study data is part of the CAPS Consortium Registry, an International registry for people screened for pancreas cancer.

REFERENCES:
- [Derived] Eshleman JR, Norris AL, Sadakari Y, Debeljak M, Borges M, Harrington C, Lin E, Brant A, Barkley T, Almario JA, Topazian M, Farrell J, Syngal S, Lee JH, Yu J, Hruban RH, Kanda M, Canto MI, Goggins M. KRAS and guanine nucleotide-binding protein mutations in pancreatic juice collected from the duodenum of patients at high risk for neoplasia undergoing endoscopic ultrasound. Clin Gastroenterol Hepatol. 2015 May;13(5):963-9.e4. doi: 10.1016/j.cgh.2014.11.028. Epub 2014 Dec 4. PMID 25481712
- [Derived] Kanda M, Sadakari Y, Borges M, Topazian M, Farrell J, Syngal S, Lee J, Kamel I, Lennon AM, Knight S, Fujiwara S, Hruban RH, Canto MI, Goggins M. Mutant TP53 in duodenal samples of pancreatic juice from patients with pancreatic cancer or high-grade dysplasia. Clin Gastroenterol Hepatol. 2013 Jun;11(6):719-30.e5. doi: 10.1016/j.cgh.2012.11.016. Epub 2012 Nov 28. PMID 23200980